CLINICAL TRIAL: NCT05955586
Title: A Phase 1, Single-center, Open-label Study to Assess the Intrapulmonary Pharmacokinetics of SPR719 by Comparing the Plasma, Epithelial Lining Fluid, and Alveolar Macrophage Concentrations Following the Oral Administration of Multiple Doses of SPR720 in Healthy Volunteers.
Brief Title: A Study to Assess the Intrapulmonary Pharmacokinetics (PK) of SPR719 by Comparing the Plasma, Epithelial Lining Fluid, and Alveolar Macrophage Concentrations Following the Oral Administration of Multiple Doses of SPR720 in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPR720-103
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPR720 (Experimental): Healthy participants will receive SPR720 1000 mg capsule, orally, for 7 days.
  Interventions: Drug: SPR720

INTERVENTIONS:
Drug: SPR720 — SPR720 1000 mg (250 mg*4 capsules) will be administered orally.

SUMMARY:
The primary purpose of this study is to evaluate the intrapulmonary PK, including epithelial lining fluid (ELF) and alveolar macrophages (AM) concentrations, of SPR719 compared to plasma concentrations of SPR719 (the active moiety in plasma of the prodrug SPR720) after oral administration of SPR720 1000 milligram (mg) capsules every 24 hours for 7 consecutive doses.

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index (BMI) ≥18.0 and ≤32.0 kilograms per meter square (kg/m^2) and weight between 55.0 and 100.0 kilograms (kg) (inclusive).
2. Forced expiratory volume in 1 second (FEV1) of at least 80% of predicted value at screening visit.
3. Have suitable venous access for blood sampling.
4. Ability and willingness to abstain from alcohol, caffeine, xanthine-containing beverages or food or product containing any of these from 48 hours prior to study drug administration until discharge from the clinical research unit (CRU).

Key Exclusion Criteria:

1. History of clinically significant acute illness or surgery within the previous 3 months prior to Screening Visit or Day -1.
2. Known history of clinically significant hypersensitivity reaction or anaphylaxis to SPR720 or an aminobenzimidazole.
3. Any condition possibly affecting drug absorption (e.g. previous surgery on the gastrointestinal tract [including removal of parts of the stomach, bowel, liver, gall bladder, or pancreas]).
4. Participants who are unable to demonstrate the ability to swallow the dosage forms.
5. Receipt of any other investigational medicinal product or participation in another investigational clinical study that included drug treatment within 30 days prior to Day 1 dose (based on the timing of the last Follow-up Visit in the previous study to Day 1 of the current study).

NOTE: Other inclusion and exclusion criteria as per protocol may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve from Time Zero to 24 Hours (AUC0-24) of SPR719 in plasma, ELF and AM | Predose on Day 6 and post-dose at multiple time points up to Day 8
Maximum Observed Concentration (Cmax) of SPR719 in plasma, ELF and AM | Predose on Day 6 and post-dose at multiple time points up to Day 8
Time to the Maximum Observed Concentration (Tmax) of SPR719 in plasma, ELF and AM | Predose on Day 6 and post-dose at multiple time points up to Day 8

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From first dose of study drug until the follow-up visit (up to 15 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Associates, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodvold KA, Gotfried MH, Ussery XT, Wong SL, Hamed KA. Intrapulmonary pharmacokinetics of SPR719 following oral administration of SPR720 to healthy volunteers. Antimicrob Agents Chemother. 2024 Nov 6;68(11):e0110324. doi: 10.1128/aac.01103-24. Epub 2024 Oct 1. PMID 39352135